CLINICAL TRIAL: NCT00888134
Title: Phase II Clinical Trial of the MEK 1/2 Inhibitor AZD6244 in Cancers With BRAF Mutations Identified by Prospective Genotypic Analysis
Brief Title: Selumetinib in Cancers With BRAF Mutations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00576; NCI-2013-00576 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA006516 (NIH); U01CA062490 (NIH); CDR642346; N01CM62206 (NIH); 09-005 (Other: Massachusetts General Hospital Cancer Center); 8281 (Other: CTEP)
Record Dates: First submitted 2009-04-23; First posted 2009-04-27 (Estimated); Results first posted 2016-01-15 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2015-07

CONDITIONS: Adult Solid Neoplasm
MeSH Terms: interventions — AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (selumetinib) (Experimental): Patients receive selumetinib PO BID for 3 weeks. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Selumetinib

INTERVENTIONS:
Drug: Selumetinib — Given PO
  Other Names: ARRY-142886; AZD6244; MEK Inhibitor AZD6244

SUMMARY:
The purpose of this research study is to determine if selumetinib is safe and effective in treating patients with cancers with a mutated BRAF gene. Selumetinib is an investigational drug that works by blocking a protein called MEK, which is known to play a role in the growth of cancer cells lines and tumors that have a mutated BRAF gene. There are multiple types of cancers that have mutations in the BRAF gene and depend on the activity of this gene for their growth and survival.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the objective response rate to AZD6244 (selumetinib) in patients with cancers other than melanoma in which BRAF mutations have been identified prospectively.

SECONDARY OBJECTIVES:

I. To evaluate progression-free survival in subjects treated with AZD6244. II. To obtain a preliminary estimate of the objective response rate in non-small cell lung cancers and colon cancers with BRAF mutations.

III. To explore biologic correlates of responsiveness to AZD6244, and specifically to correlate AKT pathway activity with sensitivity to MEK inhibition in the BRAF mutant class of tumors.

IV. To estimate the sensitivity and specificity of detection of the BRAF V600E mutation in circulating tumor cells (CTC) using a microfluidic platform (the 'CTC-chip').

OUTLINE:

Patients receive selumetinib orally (PO) twice daily (BID) for 3 weeks. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 6 months for 1 year, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign a written informed consent document
* Histologically confirmed metastatic or unresectable solid tumor
* Results from tumor tissue analysis that show a glutamic acid-for-valine substitution at amino acid position 600 in the BRAF gene (V600E) or other activating BRAF mutation, as determined by high-throughput genotyping
* Patients may have received any number of prior systemic treatments for their cancer
* At least one measurable site of disease by CT, according to standard RECIST criteria 1.0
* ECOG performance status 0-1
* Absolute neutrophil count > 1500 per cubic mm
* Platelet count > 100,000 per cubic mm
* Hemoglobin > 9 g/dl
* Serum bilirubin < 1.5 x upper limit of normal
* Serum AST and ALT < 2.5 x upper limit of normal (=< 5 x upper limit of normal, for liver metastases)
* Serum creatinine < 1.5 x upper limit of normal
* For women of childbearing potential, negative serum pregnancy test and use of physician-approved method of birth control throughout the study

Exclusion Criteria:

* Estimated life expectancy > 12 weeks
* Patients with melanoma
* Have received chemotherapy or radiotherapy within 4 weeks prior to entering the study (6 weeks for nitrosoureas or mitomycin C), or a targeted therapy within 2 weeks prior to entering the study
* Have not recovered from adverse events due to agents previously administered (CTCAE v3 grade 1 or baseline)
* Currently receiving other investigational agents
* Known brain metastases, unless treated and stable off of corticosteroids for at least four weeks
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD6244
* Prior treatment with a selective inhibitor of RAF or MEK (e.g., RAF265); (note: prior sorafenib is allowed)
* Uncontrolled intercurrent illness, including but not limited to:

  * Clinically significant active infection
  * Symptomatic congestive heart failure, unstable angina pectoris, and/or cardiac arrhythmia other than atrial fibrillation
  * Psychiatric illness/social situations that would limit compliance with study requirements
* Refractory nausea or vomiting, swallowing disorder, or malabsorption syndrome that would interfere with swallowing or absorbing the study medication
* Pregnant and/or breast-feeding women
* Previous or concurrent malignancy, except for the following circumstances:

  * Disease-free for at least three years and deemed by investigator to be at low risk for recurrence of that malignancy
  * Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin)
* History of solid organ transplantation or other condition requiring the use of immunosuppressive medications
* Uncontrolled hypertension (systolic BP >= 150 or diastolic BP >= 100 that cannot be controlled with medications)
* A mean left ventricular ejection fraction (LVEF) less than 45%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Lawrence, Principal Investigator — Massachusetts General Hospital
Locations (5):
- United States (5):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants 'complete' the treatment period if they ended their treatment for disease progression, unacceptable toxicity, withdrawal of consent, or intercurrent illness. Those participants who completed treatment then enter a follow-up period when they are followed until death or lost-to-follow-up.
Groups:
- Treatment (Selumetinib): Patients receive selumetinib PO BID for 3 weeks. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Selumetinib: Given PO
Period: Treatment With Study Drug
Arm/Group | Treatment (Selumetinib)
Started | 28
Completed | 27 (21 had progressive disease; 5 had unacceptable toxicity; 1 finished treatment)
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Follow-up
Arm/Group | Treatment (Selumetinib)
Started | 27
Completed | 26 (23 died; 3 were lost-to-follow-up)
Not Completed | 1
Not completed — being followed for long-term survival | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Selumetinib)
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 28
Type of cancer [Number; unit: participants]
  Non small-cell lung cancer | 14
  Colon cancer | 10
  Other cancer | 4

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate in Patients With Cancers Other Than Melanoma
Description: Percentage of participants achieving either complete response (disappearance of all target lesions) or partial response (at least a 30% decrease in the sum of the longest diameter of target lesions, when compared with baseline) using CT (computed tomography) scans (which are done every 6 weeks).
Time Frame: 4 years
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Selumetinib)
Number analyzed (Participants) | 28
percentage of participants | 0

2. Secondary Outcome: AKT Pathway Activity
Description: Correlation between response to AZD6244 and mutational analysis of AKT pathway (an intracellular signaling pathway important in regulating the cell cycle)
Time Frame: Up to 4 years
Population: Samples and data were not collected for this outcome.
Arm/Group | Treatment (Selumetinib)
Number analyzed (Participants) | 0

3. Secondary Outcome: Objective Response Rate in Patients With Non-small Cell Lung Cancers and Colon Cancers
Description: Percentage of participants with either colon cancer or non-small cell lung cancer achieving either complete response (disappearance of all target lesions) or partial response (at least a 30% decrease in the sum of the longest diameter of target lesions, when compared with baseline) using CT (computed tomography) scans.
Time Frame: Up to 4 years
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Selumetinib)
Number analyzed (Participants) | 24
percentage of participants | 0

4. Secondary Outcome: Progression-free Survival
Description: Reported as percentage of participants alive and progression free at 4-months. Will be estimated using Kaplan-Meier survival curves. Confidence intervals will be calculated and reported.
Time Frame: 4 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Selumetinib)
Number analyzed (Participants) | 28
percentage of participants | 21.4 [8.7 to 37.8]

5. Secondary Outcome: Sensitivity and Specificity of Detection of the BRAF V600E Mutation in CTC Using the CTC-chip
Time Frame: Up to 4 years
Population: Samples and data were not collected for this outcome.
Arm/Group | Treatment (Selumetinib)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events experienced by participants will be followed for 30 days after participant stops treatment. (if ongoing beyond 30 days, they were contacted by the study team until the event resolved)
Description: Participants were seen every 3 weeks during study treatment for physical exam, vital signs and laboratory assessments.
Arm/Group | Treatment (Selumetinib)
Serious Adverse Events (participants affected / at risk) | 17/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Selumetinib) (N=28)
hypothyroidism (Endocrine disorders) | 1
SGPT (Metabolism and nutrition disorders) | 3
Fistula (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
pulmonary / URT infection (Infections and infestations) | 1
malignant ascites (Gastrointestinal disorders) | 1
ileus (Gastrointestinal disorders) | 1
SGOT (Metabolism and nutrition disorders) | 1
confusion (Psychiatric disorders) | 1
fatigue (General disorders) | 1
mental status changes (Psychiatric disorders) | 1
fatal progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
increased intraocular pressure (Eye disorders) | 1
dry skin (Skin and subcutaneous tissue disorders) | 1
blurry vision (Eye disorders) | 2
skin infection (Skin and subcutaneous tissue disorders) | 2
joint pain (Musculoskeletal and connective tissue disorders) | 1
muscle pain (Musculoskeletal and connective tissue disorders) | 1
hypoalbuminemia (Metabolism and nutrition disorders) | 1
retinopathy (Eye disorders) | 1
dizziness (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Selumetinib) (N=28)
allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
tinnitus (Ear and labyrinth disorders) | 2
hemoglobin - low (Blood and lymphatic system disorders) | 19
leukocytes (Blood and lymphatic system disorders) | 2
lymphopenia (Blood and lymphatic system disorders) | 8
platelets (Blood and lymphatic system disorders) | 6
hypertension (Cardiac disorders) | 3
INR (Investigations) | 3
PTT (Investigations) | 3
fatigue (General disorders) | 19
fever (without neutropenia) (General disorders) | 2
insomnia (Psychiatric disorders) | 5
dry skin (Skin and subcutaneous tissue disorders) | 3
nail changes (Skin and subcutaneous tissue disorders) | 3
pruritis (Skin and subcutaneous tissue disorders) | 4
rash/desquamation (Skin and subcutaneous tissue disorders) | 6
rash: acneiform (Skin and subcutaneous tissue disorders) | 19
rash: erythema multiforme (Skin and subcutaneous tissue disorders) | 2
skin - other (Skin and subcutaneous tissue disorders) | 4
anorexia (Gastrointestinal disorders) | 5
constipation (Gastrointestinal disorders) | 8
diarrhea (Gastrointestinal disorders) | 14
dry mouth (Gastrointestinal disorders) | 3
fistula (Gastrointestinal disorders) | 2
mucositis (Gastrointestinal disorders) | 4
nausea (Gastrointestinal disorders) | 15
taste disturbance (Gastrointestinal disorders) | 2
vomiting (Gastrointestinal disorders) | 13
hemorrhage - anus (Gastrointestinal disorders) | 2
hemorrhage - nose (Respiratory, thoracic and mediastinal disorders) | 2
edema - head and neck (Blood and lymphatic system disorders) | 5
edema - limb (Blood and lymphatic system disorders) | 14
edema - trunk (Blood and lymphatic system disorders) | 2
hypoalbuminemia (Metabolism and nutrition disorders) | 16
alkaline phosphatase (Metabolism and nutrition disorders) | 17
SGPT (Metabolism and nutrition disorders) | 10
SGOT (Metabolism and nutrition disorders) | 21
bicarbonate (Metabolism and nutrition disorders) | 4
bilirubin (Metabolism and nutrition disorders) | 3
hypocalcemia (Metabolism and nutrition disorders) | 7
hypercholesterolemia (Metabolism and nutrition disorders) | 2
creatinine (Metabolism and nutrition disorders) | 3
hyperglycemia (Metabolism and nutrition disorders) | 20
hypoglycemia (Metabolism and nutrition disorders) | 2
hypermagnesemia (Metabolism and nutrition disorders) | 3
hypomagnesemia (Metabolism and nutrition disorders) | 8
hypophosphatemia (Metabolism and nutrition disorders) | 3
hyperkalemia (Metabolism and nutrition disorders) | 6
hypokalemia (Metabolism and nutrition disorders) | 7
hyponatremia (Metabolism and nutrition disorders) | 8
dizziness (Nervous system disorders) | 6
depression (Psychiatric disorders) | 4
neuropathy - sensory (Nervous system disorders) | 7
tearing (Eye disorders) | 2
abdominal pain (Gastrointestinal disorders) | 8
back pain (Musculoskeletal and connective tissue disorders) | 7
extremity - limb pain (Musculoskeletal and connective tissue disorders) | 3
headache (Nervous system disorders) | 3
joint pain (Musculoskeletal and connective tissue disorders) | 2
cough (Respiratory, thoracic and mediastinal disorders) | 13
dyspnea (Respiratory, thoracic and mediastinal disorders) | 10
voice changes/ dysarthria (Respiratory, thoracic and mediastinal disorders) | 4
infection (Infections and infestations) | 5
other (Skin and subcutaneous tissue disorders) | 4 — AEs not falling into pre-defined CTCAE categories
other (Gastrointestinal disorders) | 3 — AEs not falling into CTCAE categories
other (Metabolism and nutrition disorders) | 5 — AEs not falling into CTCAE categories
other (Eye disorders) | 3 — AEs not falling into CTCAE categories
other (Respiratory, thoracic and mediastinal disorders) | 4 — AEs not falling into CTCAE categories

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less